CLINICAL TRIAL: NCT06724419
Title: Efficacy of Nutrition Education in Alleviating Premenstrual Syndrome (PMS) Among Chinese College Students at Hainan University, China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Foo Chai Nien, Assistant Professor, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: U/SERC/56(A)-432/2024
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Premenstrual Syndrome-PMS
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The nutrition education-based intervention program will span 6 weeks, providing participants with comprehensive nutrition education based on dietary guidelines and comprising 8 topics , each lasting approximately 60-120 minutes. The aim is to comprehensively promote participants' adoption of a healthy lifestyle through various educational interventions, and each participant will be provided with the PMS management booklet.
  Interventions: Behavioral: Nutrition education-based intervention
- Control group (No Intervention): The participants in the "passive" control group will receive no further intervention and will each be provided with The PMS Management Booklet.

INTERVENTIONS:
Behavioral: Nutrition education-based intervention — The nutrition education-based intervention program will span 6 weeks, providing participants with comprehensive nutrition education based on dietary guidelines and comprising 8 topics , each lasting approximately 60-120 minutes.The aim is to comprehensively promote participants' adoption of a healthy lifestyle through various educational interventions, and each participant will be provided with the PMS management booklet.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the efficacy of nutrition education-based intervention on PMS severity, perceived stress, and lifestyle-related outcomes among the students at Hainan Vocational University of Science and Technology

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS), occurring during the luteal phase of the menstrual cycle and spontaneously resolving after menstruation begins, is a prevalent psychological and somatic disorder among women of reproductive age.Lifestyle modifications can help alleviate PMS symptoms, including dietary changes (such as reducing salt and sugar intake or increasing consumption of vegetables and fruits), engaging in regular physical activity, stress management, and avoiding smoking.This study is a parallel, unblinded, randomized controlled trial assessing the efficacy of nutrition education-based intervention on PMS severity, perceived stress, and lifestyle-related outcomes in Chinese college students. Participants will be randomly assigned to two groups: the nutrition education-based intervention group (NEI) and the control group. The nutrition education-based intervention program will span 6 weeks. The participants in the "passive" control group will receive no further intervention and will each be provided with The PMS Management Booklet. Data will be collected through online surveys at baseline, post-intervention, and at 1-month and 3-month follow-up points after the completion of the intervention. Data analysis will be performed using SPSS 26.0.

ELIGIBILITY:
Inclusion Criteria:

1. Females students aged 18 to 30 years
2. PMS scores（6-36）
3. Regular menstrual cycles (defined as a menstrual cycle of 21 to 35 days)
4. Not using hormonal compounds (such as contraceptive pills), drugs (such as fluoxetine and escitalopram), or non-drug treatments affecting premenstrual syndrome, such as special diets
5. No participation in interventional studies related to premenstrual syndrome in the past 6 months

Exclusion Criteria:

1. Amenorrhea
2. Polycystic ovarian disease (PCOD)
3. Those who are unable to attend according to intervention protocol

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
premenstrual syndrome severity | Baseline, Immediate post, after 1 month and 3 months after Intervention
  Premenstrual Syndrome Scale (PMSS):
  A total score of 6-10 on the questionnaire indicated mild PMS, 11-20 indicated moderate PMS, and more than 20 indicated severe PMS.

SECONDARY OUTCOMES:
Perceived Stress | Baseline, Immediate post, after 1 month and 3 months after Intervention
  Perceived Stress Scale (PSS):
  Low stress (0-13), moderate stress (14-26), and high stress (27-40)
physical activity | Baseline, Immediate post, after 1 month and 3 months after Intervention
  International physical activity questionnaire-short form (IPAQ-SF) ;MET-minutes/week will be used as a measure of the volume of activity. Total physical activity MET-minutes/week will be calculated as the sum of Walking + Moderate + Vigorous MET-minutes/week scores.
Dietary intake quality | Baseline, Immediate post, after 1 month and 3 months after Intervention
  Chinese Healthy Eating Index (CHEI);The total score, ranging from 0 to 100, summarizes all 17 components, with a higher score indicating better diet quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan Vocational University of Science and Technology, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No